CLINICAL TRIAL: NCT05952401
Title: Implementation Science to Reduce the Disparity in Tobacco Treatment Among Individuals With Serious Mental Illness (ISRAISE)
Brief Title: Implementation Science to Reduce the Disparity in Tobacco Treatment Among Individuals With Serious Mental Illness
Acronym: ISRAISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202307051; P50CA244431 (NIH)
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Results first posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Smoking; Smoking Cessation; Tobacco Use Cessation
Keywords: Patient Reported Outcomes; Smoking Cessation; Smoking Behaviors; Nicotine Addiction; Tobacco treatment
MeSH Terms: conditions — Smoking; Smoking Cessation; Tobacco Use Cessation; Tobacco Use Disorder

STUDY DESIGN:
Intervention Model Description: Patients will be randomized on a 1:1 basis to usual care or intervention 'nudges to quit'.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Patients will receive general brief advice about smoking cessation at patient tobacco treatment needs assessment then receive the intervention at 3 months.
  Interventions: Behavioral: Usual Care
- "Nudges to Quit" (Experimental): Patients will receive a multilevel intervention that includes reminders to care team to increase tobacco treatment engagement.
  Interventions: Behavioral: "Nudges"

INTERVENTIONS:
Behavioral: Usual Care — Usual care will be informed by practice guidelines (patient smoking cessation handout and brief advice).
  Arms: Usual Care
Behavioral: "Nudges" — Patients in the experimental arm will receive practice guidelines (patient smoking cessation handout and brief advice) and "Nudges to Quit", guideline-informed messages immediately following patient tobacco treatment needs assessment.
  Arms: "Nudges to Quit"

SUMMARY:
This is a pilot trial to examine the feasibility and preliminary effect of a multilevel intervention 'Nudges to Quit' on smoking cessation in patients with serious mental illness who smoke in a community mental health center (CMHC). "Nudges to Quit" is a multilevel intervention to increate engagement of patient, case worker, and pharmacist with tobacco treatment. The pilot trial is to generate the needed evidence for designing a future large trial to evaluate the effect of 'Nudges to Quit' as a multilevel intervention to increase tobacco treatment and reduce tobacco use among patients with serious mental illness.

DETAILED DESCRIPTION:
The overarching goal of this pilot project is to reduce the disparity in the treatment of tobacco use among individuals with serious mental illness (SMI) with low burden, multi-level implementation strategies, an important need reflected in existing evidence and a recent survey of community needs. Individuals with SMI have a much higher smoking prevalence (60% vs. 15%) and die 25 years earlier compared to the general population. Despite the fact that SMI patients express interest in and have success with evidence-based smoking cessation treatment, inadequate provision of treatment in community mental health centers (CMHCs) contributes to the high smoking prevalence and related health consequences among the mentally ill. The pilot trial aims to understand the feasibility and preliminary effects of a multilevel intervention "Nudges to Quit," designed to increase patient, case worker, and pharmacist engagement with tobacco treatment in a community mental health clinic setting. Therefore, the investigators propose a pilot randomized trial of 60 patients. Patients will be randomized with 1:1 allocation to usual care vs. intervention "Nudges to Quit". All patients will receive pre-appointment tobacco treatment needs assessment (t1) with patient input as decision support for their care team. For patients in the intervention arm, their care team (case worker and pharmacist) will receive nudge reminders based on patient-reported tobacco treatment need assessment to offer tobacco treatment. For patients in the usual care arm, the team will proceed with usual care and receive the intervention at 3 months post-enrollment (t2) to ensure all participants will receive benefit from the intervention with variation in timing. All patients will receive a baseline (t1), 3 month (t2), and 6 month follow-up survey (t3). In Aim 1, the investigators will test the effect of nudges on patient receipt of tobacco treatment. The investigators hypothesize patient receipt of tobacco cessation treatment such as medication and counseling will be higher after delivery of nudges over usual care. In Aim 2, the investigators will test the effect of nudges on smoking behaviors. The investigators hypothesize smoking behaviors will be positively effected in the nudges to quit group compared to usual care. In Aim 3, the investigators will evaluate the feasibility and preliminary effect of this pilot project for a future R01 proposal to systematically evaluate this multilevel intervention adapted for CMHCs.

ELIGIBILITY:
Inclusion Criteria:

* Patient of participating clinic
* Current smoker, >5 cigarettes per day
* Age 18 years or older
* Can speak and understand English

Exclusion Criteria:

* Active use or receipt of tobacco treatment (medication or counseling) within the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2025-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Li-Shiun Chen, M.D., MPH, ScD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 02/02/2024 and closed to participant enrollment on 09/27/2024.
Pre-assignment Details: The study consented 73 participants and 14 were excluded after consenting due to loss of contact or not meeting all eligibility criteria prior to randomization. 59 were considered enrolled and 14 were not considered enrolled in the study per the policy of the institution.
Period: Overall Study
Arm/Group | Usual Care | "Nudges to Quit"
Started | 30 | 29
Completed | 26 | 28
Not Completed | 4 | 1
Not completed — Lost to Follow-up | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | "Nudges to Quit" | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Customized [Count of Participants; unit: Participants]
  24-40 years | 6 | 10 | 16
  41-46 years | 11 | 3 | 14
  47-59 years | 5 | 9 | 14
  60-72 years | 8 | 7 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 31
  Male | 13 | 15 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 28 | 27 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 11 | 27
  White | 12 | 14 | 26
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 30 | 29 | 59

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Receiving Any Tobacco Treatment
Description: This will be quantified by the proportion of patients who receive any tobacco treatment (medication and/or counseling).
Time Frame: At 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | "Nudges to Quit"
Number analyzed (Participants) | 30 | 29
Participants
  Received treatment | 18 | 23
  Did not receive treatment | 12 | 6

2. Secondary Outcome: Proportion of Patients Receiving Any Tobacco Treatment
Description: This will be quantified by the proportion of patients who receive any tobacco treatment (medication and/or counseling).
Time Frame: At 6 months
Reporting Status: Not Posted

3. Secondary Outcome: Readiness to Quit Smoking
Description: This will be quantified by the proportion of current smokers in the stage of change classifications of Precontemplation, Contemplation, Preparation, or Action.
Time Frame: At 3 months, 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Smoking Abstinence
Description: This will be quantified by the proportion of smokers with bioverified point prevalence abstinence smoking abstinence at 3 months.
Time Frame: 3 months post intervention
Population: 5 participants from the Usual Care arm and 3 participants from the "Nudges to Quit" arm are not included because the participants did not complete the 3-month assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | "Nudges to Quit"
Number analyzed (Participants) | 25 | 26
Participants
  Achieved Smoking Abstinence (<5ppm) | 0 | 0
  Self-Reported Smoking Abstinence, but did not Achieve Bioverified Smoking Abstinence (<5ppm) | 3 | 0
  Did not Self-Report Smoking Abstinence and did not Achieve Bioverified Smoking Abstinence (<5ppm) | 22 | 26

5. Secondary Outcome: Abstinence Outcomes Across Multiple Time Points
Description: The outcome measure is abstinence (self-reported no smoking (not even a puff of a cigarette) for at least seven days prior to the assessment) over these time points.
Time Frame: At 3 months, 6 months
Reporting Status: Not Posted

6. Secondary Outcome: Smoking Quantity Across Multiple Time Points
Description: The outcome measure is smoking quantity (self-reported average cigarettes smoked per day for the past 30 days prior to the assessment) over these time points.
Time Frame: At 3 months, 6 months
Reporting Status: Not Posted

7. Secondary Outcome: Quit Attempts
Description: This outcome measure is the number of quit attempts over these time points.
Time Frame: At 3 months, 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months (07/01/2024 - 12/31/2024)
Description: As part of this study, no participants experienced all-cause mortality or any serious adverse events
Arm/Group | Usual Care | "Nudges to Quit"
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 0/30 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-22): https://cdn.clinicaltrials.gov/large-docs/01/NCT05952401/Prot_SAP_000.pdf
  • Informed Consent Form (2025-01-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT05952401/ICF_001.pdf